CLINICAL TRIAL: NCT04391374
Title: The Role of Hemostatic Markers of Endothelial Dysfunction in the Development of Disease Progression, Thrombotic Complications and Restenosis in Patients With Atherosclerotic Peripheral Artery Disease
Brief Title: Hemostatic Endothelial Dysfunction in Patients With Peripheral Artery Disease
Status: Completed | Type: Observational
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 05/18
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Artery Disease; Restenosis of Peripheral Vascular Stent; Restenosis, Vascular Graft; Endothelial Dysfunction
Keywords: hemostasis, endothelial dysfunction, restenosis, thrombosis
MeSH Terms: conditions — Peripheral Arterial Disease; Graft Occlusion, Vascular; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood samples for the assessment of the concentration of NO metabolites, PAI-1, sEPCR, and activity of vWF, FVIII.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conservative treatment: Subjects with atherosclerotic peripheral artery disease (PAD) who undergo standard of care conservative treatment according to the current PAD guidelines.
- Peripheral artery bypass grafting: Subjects with atherosclerotic peripheral artery disease who undergo an open bypass grafting with synthetic prosthesis in aorto-iliac or femoro-popliteal position
  Interventions: Procedure: an arterial reconstructive procedure
- Peripheral artery balloon angioplasty and stenting: Subjects with atherosclerotic peripheral artery disease who undergo endovascular balloon angioplasty and stenting with bare-metal stents in aorto-iliac or femoro-popliteal position
  Interventions: Procedure: an arterial reconstructive procedure

INTERVENTIONS:
Procedure: an arterial reconstructive procedure
  Groups: Peripheral artery balloon angioplasty and stenting; Peripheral artery bypass grafting

SUMMARY:
The study is aimed at evaluating the role of the activity of the key hemostatic parameters of endothelial dysfunction (nitric oxide II (NO) metabolites, plasmin activator inhibitor-1 (PAI-1), von Willebrand factor (vWF), coagulation factor VIII (FVIII), soluble endothelial protein C receptors (sEPCR)) in the development of disease progression, thrombotic complications and restenosis in subjects with atherosclerotic peripheral artery disease.

DETAILED DESCRIPTION:
The study will involve patients with atherosclerotic peripheral artery disease (Rutherford category 3-5). The subjects are to be divided into three groups:

Group A: patients who undergo bypass surgery with a synthetic graft on aorto-iliac or femoro-popliteal segment; Group B: patients who undergo endovascular balloon angioplasty and stenting on aorto-iliac or femoro-popliteal segment; Group C: patients who undergo standard of care conservative treatment.

Decisions on revascularization or conservative treatment alone is to be made by a team of vascular specialists in accordance with the severity of the disease, previous treatment, anatomy, possible need for repeat procedures in the future, and patient's preferences.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females older than 40 years of age;
2. Presence of peripheral arterial disease of atherosclerotic origin.

Exclusion Criteria:

1. Males or females younger than 40 years of age;
2. Chronic lower limb ischemia of other ethiology (Buerger's disease, aortoarteritis etc.);
3. Active cancer or remission period less than 5 years;
4. Decompensated diabetes mellitus;
5. Pregnancy or breast-feeding for females.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective study is aimed at enrolling 200 patients with atherosclerotic peripheral arterial disease, Rutherford category 3-5. The patients with PAD are scheduled to undergo either open or endovascular reconstructive procedures on aorto-iliac and femoro-popliteal segment or conservative treatment alone. The subjects of similar age, sex, and ethnicity are to be divided into three groups, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
thrombosis | 1 year
  incidence of thrombotic complications in the target arterial segment
restenosis | 1 year
  incidence of restenosis in the target arterial segment
progression of atherosclerosis | 1 year
  detection of newly formed or progressing peripheral atherosclerotic lesions

SECONDARY OUTCOMES:
limb salvage rate | 1 year
  limb salvage rate in the target extremity
acute myocardial infarction | 1 year
  incidence of acute myocardial infarction
mortality rate | 1 year
  overall mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Nina Mzhavanadze, MD, PhD, Principal Investigator — RyazSMU

IPD SHARING:
Plan to Share IPD: Undecided
Basic demographic data, including sex, age, and ethnicity are to be shared if allowed by the privacy policy.

REFERENCES:
- [Result] Kalinin RE, Suchkov IA, Mzhavanadze ND, Zhurina ON, Klimentova EA, Povarov VO. Coagulation Factor Activity and Hemostatic Markers of Endothelial Dysfunction in Patients with Peripheral Arterial Disease. Vasc Specialist Int. 2021 Aug 5;37:26. doi: 10.5758/vsi.210010. PMID 34349046
- [Result] Kalinin RE, Suchkov IA, Mzhavanadze ND, Demikhov VG, Zhurina ON, Klimentova EA. [Hemostatic changes in patients with peripheral artery disease before and after bypass surgery]. Khirurgiia (Mosk). 2018;(8):46-49. doi: 10.17116/hirurgia2018846. Russian. PMID 30113592